CLINICAL TRIAL: NCT05135741
Title: Role of Pressure Bio Feedback in Management of Forward Head Posture for Computer Users at BUMDC
Acronym: BUMDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahria University (Other)
Responsible Party: Principal Investigator, Rabia Khan, Lecturer\Clinical Instructor, Bahria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERC 12/2020
Record Dates: First submitted 2021-11-03; First posted 2021-11-26 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Forward Head Posture
Keywords: Bio Feedback; Deep Cervical Flexor; Neck pain; Forward head posture; Neck Disability Index
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pressure bio feedback (Experimental): Experimental
  Interventions: Device: pressure bio feedback
- deep cervical exercises (Experimental): comparative
  Interventions: Device: pressure bio feedback

INTERVENTIONS:
Device: pressure bio feedback — The pressure biofeedback unit was placed between the plinth and the posterior aspect of the neck just below the occiput and inflated to a baseline of 20 mmHg. A trained physiotherapist was observing and correcting any substitution movements to ensure that all subjects could perform the exercises correctly. All exercise protocols and programs were taken from previously published studies8-10. A conventional DCF exercise protocol was performed three times a week for four weeks in both groups. The duration of the conventional DCF exercise protocol was 20-30 minutes, once a day in the control group, and 15-20 minutes, once a day in the experimental group

SUMMARY:
Objective: The aim of present study is to explore the effectiveness of pressure bio feedback in treatment of occupational forward head posture on computer users.

DETAILED DESCRIPTION:
Material & Methods: This Randomized Control Trial was conducted in Bahria University College of Physical Therapy, Karachi. Ethical approval was prior taken from Institute Review Board. there were 32 participants selected randomly equally in experimental and control group. Both male and female were included with age of 25 to 55 years currently employees of Bahria University (BUMDC) having forward head posture or complaining neck pain were included. Exclusion was age less than 25 years, history of cervical trauma or surgery, any neurological conditions or cervical pathology. Experimental Group was given DCF exercises with Pressure Biofeedback Unit (PBU) and Control Group was given Conventional DCF Exercises. SPSS version 23.0 was used for analysis.

ELIGIBILITY:
Inclusion Criteria:

- Both male and female age of 25 to 55 currently employees of Bahria University (BUMDC) having forward head posture complaining neck pain.

Exclusion Criteria:

* Students of Bahria University history of cervical trauma or surgery any neurological conditions or cervical pathology

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
change in range of cervical flexion | 15 minutes before and after exercises for 4 weeks
  pre and post range of cervical flexion assessed through CROM device
change in range of right and left lateral rotations | 15 minutes before and after exercises for 4 weeks
  pre and post right and left lateral rotations assessed through CROM device

SECONDARY OUTCOMES:
improvement in capacity of heavy weight lifting | 4 weeks
  pre and post improvement in capacity of heavy weight lifting assessed through 6 kg dumbless
change in pain intensity | 4 weeks before exercise and 4 weeks after exercises
  pain was assesses pre and post using neck disability index (NDI)

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Khan, Msc(PT), Principal Investigator — Bahria University and Dental College
Locations (1):
- BUMDC, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No